CLINICAL TRIAL: NCT02729168
Title: A Bridging Study to Evaluate Safety of Rabies Vaccine INDIRAB® Five Doses (0.5ml) Post Exposure Administered Intramuscularly in Healthy Vietnamese Volunteer Aged From 5 Years Old
Brief Title: Safety Study of Rabies Vaccine INDIRAB® Five Doses (0.5ml) Post Exposure Administered Intramuscularly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Clinical Research and Clinical Trial Support for Vaccine and Biological Products (Other)
Collaborators: Bharat Biotech International Limited (Industry)
Responsible Party: Principal Investigator, Le Hoang San, Principal Investigator, Pasteur Institute, Ho Chi Minh City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VX-2015.01
Record Dates: First submitted 2016-03-25; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Rabies
Keywords: Rabies; Vaccine; Safety; INDIRAB; Vietnam
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human rabies vaccines (Experimental): Five doses 0.5 mL vaccine INDIRAB® on D0, D3, D7, D14, D28 using administered intramuscularly.
  Interventions: Biological: Human rabies vaccine

INTERVENTIONS:
Biological: Human rabies vaccine
  Other Names: INDIRAB®

SUMMARY:
An open label, non-comparative bridging study to evaluate the safety of Rabies vaccine INDIRAB® in Healthy Vietnamese volunteer aged from 5 years old.

DETAILED DESCRIPTION:
The trial is a bridging study to evaluate safety of Rabies vaccine INDIRAB® Five Doses (0.5 ml) post exposure administered Intramuscularly in healthy Vietnamese Volunteer Aged from 5 years old. 120 subjects will be enrolled in Cho Gao district, Tien Giang province, in which there are 100 adults (≥15 years old) and 20 children (5-<15 years old). These subjects will be received 5 doses (0.5ml) INDIRAB® on D0, 3, 7, 14 and 28.

The frequency, rate and severity of immediate adverse events (AE) within 30 minutes after vaccination, solicited and unsolicited AE within 7 days after each vaccination, the frequency and rate of serious adverse events (SAE) within 35 days after the first vaccination will be recorded as evidences for INDIRAB® safety assessment. The subjects to be included from this trial would be representative of the population of Vietnam.

The protocol has been reviewed and approved by Institutional Review Board of Pasteur Institute in Ho Chi Minh City and Vietnam Ministry of Health - Independent Ethics Committee and Vietnam Minister of Health.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female aged from 5 years old. Women of childbearing age must use an appropriate method of contraception.
2. Subjects had sign written consent form to participate in the study. With subjects aged from 5 to below 18 years old, parents/legal representative had sign written consent form for children to participate in this study.
3. Subject who gave voluntary to comply with the study requirements.

Exclusion Criteria:

1. Subjects have atopic allergy or severe allergy to any component of vaccine.
2. Subjects with mental illness, mental retardation.
3. Subjects with severe acute or chronic disease may affect safety (eg: hepatobiliary disease, kidney disease, diabetes, hypertension…).
4. Subjects received rabies vaccine.
5. Subjects with hemophilia or receiving a treatment with an anticoagulant, who are at increased risk of serious bleeding during intramuscular injection.
6. Subjects who received other vaccine within 28 days before INDIRAB® vaccination, or those who had another vaccination schedule during the study.
7. Pregnant or lactating women.
8. Subjects had been participated, are participating, are going to participate in any other clinical trials during the period of this study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety of rabies vaccine INDIRAB® by assessing the frequency, rate and severity of adverse events (local and general). | 30 minutes after vaccination
Safety of rabies vaccine INDIRAB® by assessing the frequency, rate and severity of solicited and unsolicited adverse events. | For 7 days after each vaccination
Safety of rabies vaccine INDIRAB® by assessing the frequency, rate and severity of Serious Adverse Events. | Within 35 days after the first vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Cho Gao Health Centre, Chợ Gạo, Tien Giang, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided